CLINICAL TRIAL: NCT04246996
Title: Gentamicin Intravesical Efficacy for Infection of Urinary Tract
Acronym: GIVEIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GIVEIT; 12297 (Other: Kaiser Permanente Southern California IRB); 191835 (Other: UC San Diego Health IRB)
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Urinary Tract Infection; Pelvic Organ Prolapse; Stress Urinary Incontinence
Keywords: gentamicin sulfate; pelvic organ prolapse surgery; midurethral sling; bladder instillation
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress | interventions — Gentamicins

STUDY DESIGN:
Who Masked: Participant
Masking Description: The subject will be masked as to whether she has been assigned to the gentamicin arm or the control arm. The subject will be unmasked at the completion of the 6 week follow up period.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gentamicin Arm (Active Comparator): At the completion of the subjects surgery but prior to awakening from anesthesia, 80mg of gentamicin in 50 mL of normal saline will be infused into the subject's bladder through the standard-of-care transurethral catheter by the surgeon. The surgeon will then clamp the catheter and label the catheter with the clamping time. The catheter will be clamped to prevent the gentamicin from immediately flowing out of the bladder and thus allow the gentamicin time to have an effect. The subject will then proceed as usual to the postoperative anesthesia care unit. A member of the subject's care team will unclamp the catheter after 1 hour. The subject will otherwise have usual pre-operative and post-operative care.
  Interventions: Drug: gentamicin sulfate
- Control Arm (Sham Comparator): If the patient is randomized to no instillation, at the end of the surgery but prior to awakening from anesthesia, the surgeon will clamp the catheter and label the catheter with the clamping time. The purpose of clamping the catheter for subjects receiving usual care will be to ensure patients are masked to study arm assignment if they wake up and notice their catheter. The subject will then proceed as usual to the postoperative anesthesia care unit. A member of the subject's care team will unclamp the catheter after 1 hour. The subject will otherwise have usual pre-operative and post-operative care.
  Interventions: Other: Catheter clamping only

INTERVENTIONS:
Drug: gentamicin sulfate — Subjects in the gentamicin arm will receive an bladder instillation of 80mg of gentamicin sulfate in 50 mL of normal saline through a standard-of-care Foley catheter.
  Other Names: gentamicin sulfate transurethral bladder instillation with catheter clamping for 1 hour
  Arms: Gentamicin Arm
Other: Catheter clamping only — Subjects in the control arm will have their standard-of-care transurethral catheter clamped for 1 hour post-placement to maintain subject masking to study arm.
  Arms: Control Arm

SUMMARY:
Urinary tract infection (UTI) is a common problem after surgery for pelvic organ prolapse and stress urinary incontinence. This prospective, randomized, single-masked (subject), two-parallel armed study aims to determine the effect of a single postoperative intravesical instillation of 80 mg of gentamicin sulfate in 50 mL of saline versus usual care on the proportion of women treated for UTI within 6 weeks following surgery for pelvic organ prolapse (POP) or stress urinary incontinence (SUI).

ELIGIBILITY:
Inclusion Criteria:

* Adult women undergoing pelvic organ prolapse surgery and/or stress urinary incontinence surgery with surgical plan for at least 1 cystoscopy and will leave the operating room with a standard-of-care transurethral catheter.
* Negative urine culture within 4 weeks or completion of UTI treatment ≥48 hours prior to surgery

Exclusion Criteria:

* History of allergic reaction or anaphylaxis to gentamicin sulfate or to sodium metabisulfite (one of the preservatives in the gentamicin sulfate product)
* Abnormal intraoperative urinary tract finding (e.g. bladder mass, stone, or fistula)
* Intraoperative urinary tract injury
* Suppressive recurrent UTI treatment
* Chronic indwelling catheter/self-catheterization
* Unable to provide informed consent
* Severe renal impairment - glomerular filtration rate of less than 30 mL / minute
* Current pregnancy
* Currently incarcerated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All subjects will be female because undergoing surgery for female pelvic organ prolapse and stress urinary incontinence is an inclusion criterion.
Enrollment: 370 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2021-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly L Ferrante, M.D., M.A.S., Principal Investigator — Kaiser Permanente; Marianna Alperin, M.D., M.S., Principal Investigator — UC San Diego Health
Locations (2):
- United States (2):
  - UC San Diego Health, La Jolla, California
  - Kaiser Permanente San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rieger MM, Shah NM, Ferrante KL, Tan-Kim J, Jacobs MB, Brubaker L, Alperin M. Intraoperative Gentamicin Intravesical Instillation for Prevention of Urinary Tract Infection After Urogynecologic Surgery: A Randomized Controlled Trial. Urogynecology (Phila). 2022 Dec 1;28(12):825-833. doi: 10.1097/SPV.0000000000001233. Epub 2022 Aug 23. PMID 36409639

RESULTS

PARTICIPANT FLOW:
Groups:
- Gentamicin Arm: At completion of surgery but prior to awakening from anesthesia, after ensuring the bladder is fully drained, 80mg of gentamicin in 50 mL of normal saline will be infused by the surgeon into the participants's bladder through the standard-care transurethral catheter. The surgeon will then clamp the catheter and label the catheter with the clamping time. The catheter will be clamped to prevent the gentamicin from immediately flowing out of the bladder and thus allow the gentamicin time to have an effect. The participant will then proceed as usual to the postoperative anesthesia care unit. The recovery room nurse will unclamp the catheter after 1 hour. The subject will otherwise have usual pre-operative and post-operative care.
  gentamicin sulfate: Subjects in the gentamicin arm will receive an bladder instillation of 80mg of gentamicin sulfate in 50 mL of normal saline through a standard-of-care Foley catheter.
- Control Arm: At the end of the surgery but prior to awakening from anesthesia, after ensuring the bladder is fully drained, the surgeon will clamp the catheter and label the catheter with the clamping time. The purpose of clamping the catheter for participants receiving usual care will be to ensure participants are masked to study arm assignment if they wake up and notice their catheter. The participant will then proceed as usual to the postoperative anesthesia care unit. The recovery room nurse will unclamp the catheter after 1 hour. The participant will otherwise have usual pre-operative and post-operative care.
  Catheter clamping only: Participants in the control arm will have their standard-of-care transurethral catheter clamped for 1 hour post-placement to maintain participant masking to study arm.
Period: Overall Study
Arm/Group | Gentamicin Arm | Control Arm
Started (Randomized to study arm) | 185 | 185
Completed (Analyzed) | 183 | 180
Not Completed | 2 | 5
Not completed — Physician Decision | 1 | 1
Not completed — Did not meet eligibility criteria | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gentamicin Arm | Control Arm | Total
Number analyzed (Participants) | 183 | 180 | 363
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (12.0) | 58.7 (12.8) | 58.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 180 | 363
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — As entered into electronic medical cord
  Participants
    Asian | 6 | 5 | 11
    Black | 5 | 6 | 11
    Hispanic | 70 | 61 | 131
    White Non-Hispanic | 97 | 99 | 196
    Other | 4 | 8 | 12
    Not specified | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 183 | 180 | 363
Study site [Count of Participants; unit: Participants]
  University of California San Diego | 122 | 123 | 245
  Kaiser Permanente San Diego | 61 | 57 | 118
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.5 (5.6) | 28.2 (5.1) | 28.2 (5.1)
Parity [Median (Full Range); unit: births] | 2 [0 to 8] | 2 [0 to 8] | 2 [0 to 8]
American Society of Anesthesiologists (ASA) Physical Status Classification [Median (Full Range); unit: units on a scale] — ASA 1 - A normal healthy patient, ASA 2 - A patient with mild systemic disease, ASA 3 - A patient with severe systemic disease, ASA 4 - A patient with severe systemic disease that is a constant threat to life, ASA 5 - A moribund patient who is not expected to survive without the operation, ASA 6 - A declared brain-dead patient whose organs are being removed for donor purposes
  units on a scale | 2 [1 to 4] | 2 [1 to 3] | 2 [1 to 4]
Diabetes mellitus [Count of Participants; unit: Participants] | 24 | 25 | 49
Current smoker [Count of Participants; unit: Participants] | 9 | 12 | 21
Postmenopausal [Count of Participants; unit: Participants]
  Yes | 122 | 116 | 238
  No | 47 | 48 | 95
  Unknown | 14 | 16 | 30
Current vaginal estrogen use [Count of Participants; unit: Participants] | 79 | 76 | 155
Current menopausal hormone therapy use [Count of Participants; unit: Participants] | 10 | 9 | 19
Number of culture positive UTIs in 12 months prior to surgery [Number; unit: participants]
  0 UTIs | 155 | 156 | 311
  1 UTI | 20 | 20 | 40
  2 UTIs | 6 | 3 | 9
  3 UTIs | 2 | 1 | 3
Positive urine culture within 4 weeks before surgery [Count of Participants; unit: Participants] | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Urinary Tract Infection
Description: Number of participants in each arm treated with antibiotics for urinary tract infection symptoms
Time Frame: Within 6 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Arm | Control Arm
Number analyzed (Participants) | 183 | 180
Participants | 19 | 20

2. Secondary Outcome: Adverse Events
Description: Hospital readmissions
Time Frame: Within 6 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Arm | Control Arm
Number analyzed (Participants) | 183 | 180
Participants | 5 | 6

3. Secondary Outcome: Number of Participants With Isolated Uropathogen on Post-operative Urine Culture
Time Frame: Within 6 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Arm | Control Arm
Number analyzed (Participants) | 183 | 180
Participants | 12 | 15

ADVERSE EVENTS:
Time Frame: 6 weeks after surgery
Description: Hospital readmission within 6 weeks after surgery as reported by patient or found in electronic medical record
Arm/Group | Gentamicin Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/180
Serious Adverse Events (participants affected / at risk) | 5/183 | 6/180
Other Adverse Events (participants affected / at risk) | 0/183 | 0/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gentamicin Arm (N=183) | Control Arm (N=180)
Small bowel obstruction (Gastrointestinal disorders) | 0 | 1
Reoperation for hematoma (Surgical and medical procedures) | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0
Ischemic stroke (Nervous system disorders) | 0 | 1
Diabetic Ketoacidosis (Endocrine disorders) | 0 | 1
Uncontrolled postoperative pain (Injury, poisoning and procedural complications) | 1 | 0
Acute cholecystitis (Gastrointestinal disorders) | 1 | 0
Admitted for planned breast surgery (Surgical and medical procedures) | 1 | 0
Reoperation for sling division (Renal and urinary disorders) | 0 | 1
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT04246996/Prot_SAP_000.pdf